CLINICAL TRIAL: NCT06010251
Title: Mechanisms and Utility of Multisensory Body- Representation in SCI and SCI-Related Neuropathic Pain
Brief Title: Utility of Multisensory Body-Representation in Spinal Cord Injury (SCI) With Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Eva Widerstrom-Noga, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20230447; SC220073 (Other Grant/Funding Number: CDMRP)
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries; Neuropathic Pain
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCI with pain (Experimental): Participants will undergo 2-4 weeks of combined intervention including transcranial direct current stimulation (tDCS) and bodily illusions (10 sessions total).
  Interventions: Other: tDCS and bodily illusions

INTERVENTIONS:
Other: tDCS and bodily illusions — Participants will be required to perform (in person) 10 interventions over a time frame of 2-4 weeks. They can perform this everyday or for a minimum of 2-3 times per week over 4 weeks.
  Two types of illusions will be used 15 min each, the rubber hand illusion and the walking illusion to target upper and lower limbs. These procedures will impact the body representation of the participants resulting in bodily illusions.

SUMMARY:
The purpose of this study is to investigate the effectiveness of bodily illusions combined with transcranial direct current stimulation (tDCS) on neuropathic pain symptoms and sensory functions in participants with spinal cord injury (SCI) and neuropathic pain.

ELIGIBILITY:
The study will be open to people of any ethnicity, racial background, and gender.

Inclusion criteria:

SCI with Pain:

1. Men or women
2. fluent in English
3. 18-70 years of age who have: (3a) Complete and incomplete SCI, level of injury (above L1); (3b) Persistent neuropathic pain started after the injury for a minimum of three months prior to entering the study that is at least moderate in severity, defined as ≥ 4 on a Numeric Rating Scale (NRS) ranging 0 to 10.

Exclusion criteria:

Participants will be excluded if they have:

1. Major psychiatric disease/disorder (self-reported);
2. a significant neurological trauma (self-reported) other than SCI;
3. a recent (one-year) history of alcohol or drug abuse assessed by the Drug Abuse Screening Test (DAST-10)
4. history of visual and hearing loss not corrected
5. history of epilepsy or seizures
6. any metal implants in the head, or implanted devices such as cochlea implants or cardiac pacemakers.

We will not include any special population like:

Adults unable to consent Individuals who are not yet adults (infants, children, teenagers) Pregnant women Prisoners

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Change in neuropathic pain severity assessed by Neuropathic Pain Symptom Inventory (NPSI) | Baseline, up to 4 weeks
  The NPSI is a self-reported, validated questionnaire that includes 10 items (on different pain sensations, e.g., burning, squeezing, electric-shock, etc.) used to evaluate the properties of neuropathic pain. Each item is scored on an 11-point NRS (0 meaning no symptom and 10 meaning worst symptom), with higher scores indicating more severe neuropathic pain symptoms.
Change in neuropathic pain interference assessed by pain interference questionnaire. | Baseline, up to 4 weeks
  The questionnaire consists in a numerical rating of pain interference ranging from 0= No Interference to 10=Extreme interference with activities, mood and sleep
Changes associated with sensory function/dysfunction assessed by quantitative sensory testing | Baseline, up to 4 weeks
  The sensory test assesses thermal thresholds and includes:
  cool detection threshold (CDT), warm detection threshold (WDT), cold pain threshold (CPT), hot pain threshold (HPT), all performed using the method of limits: 0 to 50 Celsius (ºC) all values will be reported in Celsius.

SECONDARY OUTCOMES:
Change in manageable pain assessed by days of manageable pain questionnaire. | Baseline, up to 4 weeks
  This item specifies the total number of days with pain during the last 7 days, including today, and the response categories ranges from 0=none to 7=seven days.
Changes of psychosocial assessed by Multidimensional Pain Inventory (pain severity subscale) | Baseline, up to 4 weeks
  Multidimensional Pain Inventory assesses the psychosocial impact of pain. This scale consists of three questions: 1) pain at the present moment; 2) pain during the past week and 3) suffering because of pain.
  The range of the responses are from 0 (no pain or suffering) to 6 (extreme pain or suffering) and the scores of these three questions will be summed to obtain a composite pain severity score.
Change in Global impression of changes by PGIC questionnaire | Baseline, up to 4 weeks
  Patients' Global Impression of Changes (PGIC) assesses patients' perceptions of changes following treatment. It is a 7-point verbal scale, with the options ranging from "very much improved" (3), "much improved" (2), "minimally improved" (1), "no change" (0), "minimally worsened" (-1) "much worsened" (-2), and "very much worsened" (-3).

CONTACTS AND LOCATIONS:
Overall Officials: Eva Widerstrom-Noga, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No